CLINICAL TRIAL: NCT05587426
Title: Postprandial Glucose, and Insulin Response of Sugars From Fiber: An Acute, Double Blind, Randomized Controlled Clinical Trial
Brief Title: A Study to Investigate the Effect of SFF on Glucose and Insulin Responses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cambridge Glycoscience (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: CG2211
Record Dates: First submitted 2022-10-17; First posted 2022-10-20 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Postprandial Glycemic Response
MeSH Terms: interventions — Glucose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Glucose - Control (Active Comparator): 20 g of glucose mixed with 250 ml of cold water
  Interventions: Dietary Supplement: Glucose
- SFF (Experimental): 20 g of SFF mixed with 250 ml of cold water
  Interventions: Dietary Supplement: SFF
- Regular chocolate chips - Control (Active Comparator): 50 g of regular chocolate chips
  Interventions: Dietary Supplement: Regular chocolate chips
- SFF chocolate chips (Experimental): 50 g of SFF chocolate chips
  Interventions: Dietary Supplement: SFF chocolate chips

INTERVENTIONS:
Dietary Supplement: SFF — Ingestion of 20g of SFF after 10-14 hours of fasting
  Arms: SFF
Dietary Supplement: Glucose — Ingestion of 20g of glucose after 10-14 hours of fasting
  Arms: Glucose - Control
Dietary Supplement: SFF chocolate chips — Ingestion of 50g of chocolate chips made with SFF after 10-14 hours of fasting
  Arms: SFF chocolate chips
Dietary Supplement: Regular chocolate chips — Ingestion of 50g of regular chocolate chips after 10-14 hours of fasting
  Arms: Regular chocolate chips - Control

SUMMARY:
This goal of this clinical study is to investigate the postprandial glycemic and insulinemic response in healthy adults after the consumption of:

1. Sugars from Fiber in comparison with dextrose
2. Sugars from Fiber incorporated into chocolate chips in comparison with regular chocolate chips

ELIGIBILITY:
Inclusion Criteria:

1. Individuals, 20-65 years of age, inclusive.
2. Body mass index (BMI) between 19 and 35 kg/m², inclusive, at screening.
3. Willing to maintain habitual diet, physical activity pattern, and body weight throughout the trial.
4. Willing to maintain current dietary supplement and non-exclusionary medication use throughout the trial.
5. Willing to avoid the consumption of alcohol, unusual food intake, and unusual physical activity 24h prior to each study visit. Failure to follow will result in rescheduled visit.
6. Understanding the study procedures and willing to provide informed consent to participate in the study and authorization to release relevant protected. health information to the study investigator.

Exclusion Criteria:

1. Failure to meet any one of the inclusion criteria.
2. Known history of gastrointestinal disease (e.g., diverticulitis, Crohns disease, coeliac disease etc.), bariatric surgery, AIDS, hepatitis, a history or presence of clinically important endocrine (including Type 1 or Type 2 diabetes mellitus), cardiovascular (including, but not limited to, atherosclerotic disease, history of myocardial infarction, peripheral arterial disease, stroke), pulmonary, or biliary diseases, or any condition which might, in the opinion of the medical director either: 1) make participation dangerous to the subject or to others, or 2) affect the results.
3. Use of medications known to influence carbohydrate metabolism, gastrointestinal function or appetite, including, but not limited to adrenergic blockers, diuretics, thiazolidinediones, metformin and systemic corticosteroids within 4 weeks of the screening visit, or any medication which might, in the opinion of the medical director either: 1) make participation dangerous to the subject or to others, or 2) affect the results.
4. Major trauma or surgical event within 3 months of screening.
5. Unwillingness or inability to comply with the experimental procedures and to follow INQUIS safety guidelines.
6. Known intolerance, sensitivity or allergy to test foods.
7. Extreme dietary habits, as judged by the Investigator (i.e. Atkins diet, very high protein diets, etc.).
8. History of cancer in the prior two years, except for non-melanoma skin cancer.
9. Exposure to any non-registered drug product within 30 d prior to screening.
10. Self-reported pregnancy or breastfeeding.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-06-03 (Actual); Primary Completion 2022-07-29 (Actual); Study Completion 2022-07-29 (Actual)

PRIMARY OUTCOMES:
Plasma glucose iAUC (T0 - T120min) after test meals | Through intervention periods of two hours
  Compare the postprandial glucose incremental area under the curve after consumption of:
  SFF compared to glucose or SFF chocolate chips compared to regular chocolate chips

SECONDARY OUTCOMES:
Plasma glucose at each time point after test meals | Through intervention periods of two hours
  Compare the postprandial glucose levels at each time point after consumption of:
  SFF compared to glucose or SFF chocolate chips compared to regular chocolate chips
Serum insulin iAUC (T0 - T120min) and each time point after test meals | Through intervention periods of two hours
  Compare the postprandial insulin levels at each time and incremental area under the curve after consumption of:
  SFF compared to glucose or SFF chocolate chips compared to regular chocolate chips

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Wolever, Ph.D, Principal Investigator — INQUIS Clinical Research
Locations (1):
- INQUIS Clinical Research, Ltd, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Moura de Oliveira Beltrame D, Simmons TJ, Jenkins AL, Dinan T, Nicholson TJ. Gastrointestinal Tolerability and Acute Glycemic Response of Oligosaccharides and Polysaccharides from Cellulose and Xylan in Healthy Adults: Two Double-Blinded, Randomized, Controlled, Cross-over Trials. J Am Nutr Assoc. 2024 May-Jun;43(4):305-314. doi: 10.1080/27697061.2023.2282615. Epub 2023 Nov 30. PMID 38032277